CLINICAL TRIAL: NCT01134393
Title: A Prospective, Open-label TElmisartan/AMlodipine Single Pill STudy to Assess the Efficacy in Patients With Essential Hypertension"..."
Brief Title: TElmisartan and AMlodipine Single Pill sTudy With Patients Not on Goal With Mono rAas Therapy-switch
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1235.33; 2009-017336-40 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Results first posted 2012-07-04 (Estimated); Last update posted 2014-01-15 (Estimated); Status verified 2013-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — telmisartan amlodipine combination

ARMS (1):
- telmisartan/amlodipine (Experimental): start low dose and uptitrate to high dose on the basis of blood pressure goal
  Interventions: Drug: telmisartan/amlodipine

INTERVENTIONS:
Drug: telmisartan/amlodipine — start low dose and uptitrate to high dose on the basis of BP goal

SUMMARY:
The general aim of this trial to determine the efficacy as measured by the percentage of patients reaching blood pressure goal at the end of the treatment period at 12 weeks. In-clinic blood pressures, home blood pressures and safety will be carefully monitored.

DETAILED DESCRIPTION:
Study Design:

ELIGIBILITY:
Inclusion criteria:

1. Ability to provide written informed consent in accordance with Good Clinical Practice and local legislation
2. Age 18 years or older
3. Patients with uncontrolled hypertension as defined SBP > 140 mmHg and SBP > 130 mmHg in patients with diabetes or renal impairment or DBP > 90 mmHg and DBP >80 mmHg in patients with diabetes or renal impairment after at least an 6 weeks of stable treatment with antihypertensive medication defined as treatment with the clinically recommended dose of a single RAAS blocking agent (Angiotensin Converting Enzym inhibition, AII Receptor Blocker and Direct Renin Inhibitor) at entering the trial. Renal impairment is defined as a creatinine >133µmol/l (1.5mg/dl) in male patients and a creatinine >124µmol/l (1.3mg/dl) in female patients or a creatinine clearance between 30-60 ml/min

Exclusion criteria:

1. Pre-menopausal women who are not surgically sterile; or are nursing or pregnant; or are not practising acceptable means of birth control or do not plan to continue using acceptable means of birth control throughout the study and do not agree to submit to pregnancy testing during participation in the trial. Acceptable methods of birth control include the transdermal patch, oral, implantable or injectable contraceptives, sexual abstinence and vasectomised partner.
2. Known or suspected secondary hypertension (e.g., renal artery stenosis or phaeochromocytoma).
3. Mean in-clinic seated cuff Systolic BP >180 mmHg and SBP >160 mmHg in patients with diabetes or renal impairment or Diastolic BP >110 mmHg and DBP >100 mmHg in patients with diabetes or renal impairment. Renal impairment is defined as a creatinine >133µmol/l (1.5mg/dl) in male patients and a creatinine >124µmol/l (1.3mg/dl) in female patients or a creatinine clearance between 30-60 ml/min.
4. Renal dysfunction as defined by the following laboratory parameters: Serum creatinine >3.0 mg/dl (or >265 ¿mol/L) and/or known creatinine clearance of <30 ml/min and/or clinical markers of severe renal impairment.
5. Bilateral renal artery stenosis, renal artery stenosis in a solitary kidney, post-renal transplant patients or patients with only one kidney.
6. Clinically relevant hypokalaemia or hyperkalaemia (i.e., <3.5 or >5.5 mEq/L).
7. Uncorrected sodium or volume depletion.
8. Primary aldosteronism.
9. Hereditary fructose intolerance.
10. Congestive heart failure New York Heart Association functional class Congestive Heart Failure III-IV (Refer to Appendix 10.1).
11. Clinically significant ventricular tachycardia, atrial fibrillation, atrial flutter or other clinically relevant cardiac arrhythmias as determined by the Investigator.
12. Biliary obstructive disorders (e.g., cholestasis) or hepatic insufficiency (defined as elevated levels of >2x bilirubin or >2x transaminases values). (Refer to Appendix 10.3)
13. Patients who have previously experienced symptoms characteristic of angioedema during treatment with ACE inhibitors or angiotensin-II receptor antagonists.
14. History of drug or alcohol dependency within six months prior to signing the informed consent form.
15. Any investigational drug therapy within one month of signing the informed consent.
16. Known hypersensitivity to any component of the trial drugs (telmisartan or amlodipine).
17. History of non-compliance or inability to comply with prescribed medications or protocol procedures.
18. Any other clinical condition which, in the opinion of the investigator, would not allow safe completion of the protocol and safe administration of the trial medication.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 502 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (47):
- Germany (10):
  - 1235.33.49010 Boehringer Ingelheim Investigational Site, Berlin
  - 1235.33.49002 Boehringer Ingelheim Investigational Site, Frankfurt
  - 1235.33.49007 Boehringer Ingelheim Investigational Site, Haag
  - 1235.33.49003 Boehringer Ingelheim Investigational Site, Heidelberg
  - 1235.33.49005 Boehringer Ingelheim Investigational Site, Künzing
  - 1235.33.49008 Boehringer Ingelheim Investigational Site, Nuremberg
  - 1235.33.49009 Boehringer Ingelheim Investigational Site, Rednitzhembach
  - 1235.33.49006 Boehringer Ingelheim Investigational Site, Rodgau-Dudenhofen
  - 1235.33.49004 Boehringer Ingelheim Investigational Site, Unterschneidheim
  - 1235.33.49001 Boehringer Ingelheim Investigational Site, Westerkappeln
- Italy (8):
  - 1235.33.39009 Boehringer Ingelheim Investigational Site, Arezzo
  - 1235.33.39002 Boehringer Ingelheim Investigational Site, Bologna
  - 1235.33.39004 Boehringer Ingelheim Investigational Site, Ferrara
  - 1235.33.39006 Boehringer Ingelheim Investigational Site, L’Aquila
  - 1235.33.39007 Boehringer Ingelheim Investigational Site, Napoli
  - 1235.33.39001 Boehringer Ingelheim Investigational Site, Pisa
  - 1235.33.39008 Boehringer Ingelheim Investigational Site, Roma
  - 1235.33.39005 Boehringer Ingelheim Investigational Site, Stradella (PV)
- Mexico (8):
  - 1235.33.52004 Boehringer Ingelheim Investigational Site, Aguascalientes
  - 1235.33.52002 Boehringer Ingelheim Investigational Site, Durango
  - 1235.33.52001 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1235.33.52003 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1235.33.52007 Boehringer Ingelheim Investigational Site, Guadalajara
  - 1235.33.52006 Boehringer Ingelheim Investigational Site, México
  - 1235.33.52009 Boehringer Ingelheim Investigational Site, México
  - 1235.33.52008 Boehringer Ingelheim Investigational Site, Monterrey
- Netherlands (9):
  - 1235.33.31007 Boehringer Ingelheim Investigational Site, 's-Hertogenbosch
  - 1235.33.31009 Boehringer Ingelheim Investigational Site, Almere Stad
  - 1235.33.31005 Boehringer Ingelheim Investigational Site, Beek en Donk
  - 1235.33.31002 Boehringer Ingelheim Investigational Site, Beerzerveld
  - 1235.33.31008 Boehringer Ingelheim Investigational Site, Ermelo
  - 1235.33.31006 Boehringer Ingelheim Investigational Site, Lichtenvoorde
  - 1235.33.31001 Boehringer Ingelheim Investigational Site, Musselkanaal
  - 1235.33.31004 Boehringer Ingelheim Investigational Site, Nijverdal
  - 1235.33.31003 Boehringer Ingelheim Investigational Site, Wildervank
- Poland (12):
  - 1235.33.48005 Boehringer Ingelheim Investigational Site, Chorzów
  - 1235.33.48002 Boehringer Ingelheim Investigational Site, Częstochowa
  - 1235.33.48003 Boehringer Ingelheim Investigational Site, Częstochowa
  - 1235.33.48010 Boehringer Ingelheim Investigational Site, Dąbrowa Górnicza
  - 1235.33.48006 Boehringer Ingelheim Investigational Site, Grodzisk Mazowiecki
  - 1235.33.48013 Boehringer Ingelheim Investigational Site, Oświęcim
  - 1235.33.48008 Boehringer Ingelheim Investigational Site, Piotrkow Trybunalski
  - 1235.33.48004 Boehringer Ingelheim Investigational Site, Poznan
  - 1235.33.48001 Boehringer Ingelheim Investigational Site, Tychy
  - 1235.33.48009 Boehringer Ingelheim Investigational Site, Tychy
  - 1235.33.48011 Boehringer Ingelheim Investigational Site, Warsaw
  - 1235.33.48007 Boehringer Ingelheim Investigational Site, Wroclaw

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This was a prospective, single-arm, open-label, uncontrolled, multi-centre, international trial. Whilst 542 patients were enrolled, 502 entered the study. Since one patient refused to take study medication, only 501 patients were treated. The Full analysis set (FAS) consisted of 494 patients and this is the basis of most data presentations.
Groups:
- T80/A5: Telmisartan 80mg plus Amlodipine 5mg fixed-dose combination
Period: Overall Study
Arm/Group | T80/A5
Started | 501 (Entered and treated.)
Completed | 449 (Completed trial medication.)
Not Completed | 52
Not completed — Adverse Event | 18
Not completed — Lack of Efficacy | 2
Not completed — Protocol Violation | 12
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 11
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Arm/Group | T80/A5
Number analyzed (Participants) | 494
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58.0 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 207
  Male | 287
Systolic Blood Pressure (SBP) at time of baseline [Mean (Standard Deviation); unit: mmHg] | 151.4 (10.2)
Diastolic Blood Pressure (DBP) at time of baseline [Mean (Standard Deviation); unit: mmHg] | 91.8 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Achieving Blood Pressure (BP) Control After 12 Weeks of Treatment Using In-clinic BP Measurements.
Description: Achieving BP control is defined as SBP<140 mmHg and DBP<90 mmHg.
Time Frame: 12 weeks
Population: Full Analysis Set (FAS) is defined as all patients who took at least one dose of trial medication, and for whom a baseline measurement and at least one post-baseline efficacy measurement were available. Last observation carried forward (LOCF) will be used.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | T80/A5
Number analyzed (Participants) | 494
Percentage of participants | 67.6 [63.3 to 71.7]

2. Secondary Outcome: BP Control After 4 and 8 Weeks of Treatment Using In-clinic BP Measurements.
Description: Achieving BP control is defined as SBP<140 mmHg and DBP<90 mmHg.
Time Frame: 4 and 8 weeks
Population: FAS and LOCF
Measure: Number; unit: Number of participants
Arm/Group | T80/A5
Number analyzed (Participants) | 494
Number of participants
  Week 4 | 262
  Week 8 | 330

3. Secondary Outcome: BP Control (Morning and Evening) After 12 Weeks of Treatment Using Home Blood Pressure Measurement (HBPM).
Description: Achieving BP control with HBPM is defined as SBP<135 mmHg and DBP<85 mmHg.
Time Frame: Week 12
Population: FAS and LOCF and with at least one post baseline HBPM measurement
Measure: Number; unit: Number of participants
Arm/Group | T80/A5
Number analyzed (Participants) | 409
Number of participants
  Morning | 179
  Evening | 172

4. Secondary Outcome: Change From Baseline Over Time in In-clinic Measured Mean SBP and Mean DBP
Time Frame: weeks 4, 8 and 12
Population: FAS with non-missing data
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | T80/A5
Number analyzed (Participants) | 494
mmHg
  Change at week 4 SBP (N=485) | -13.58 (11.95)
  Change at week 8 SBP (N=487) | -16.37 (12.34)
  Change at week 12 SBP (N=487) | -16.92 (12.24)
  Change at week 4 DBP (N=485) | -8.24 (8.77)
  Change at week 8 DBP (N=487) | -10.33 (8.88)
  Change at week 12 DBP (N=487) | -10.43 (8.83)

5. Secondary Outcome: Change From Baseline Over Time in In-clinic Measured Mean Pulse Rate
Description: Pulse pressure was not analysed for this study instead pulse rate was analysed at weeks 4, 8 and 12.
Time Frame: weeks 4, 8 and 12
Population: Treated Set (TS) with non-missing data
Measure: Mean (Standard Deviation); unit: bpm
Arm/Group | T80/A5
Number analyzed (Participants) | 501
bpm
  Change at week 4 (N=482) | 1.43 (9.22)
  Change at week 8 (N=463) | 0.32 (9.21)
  Change at week 12 (N=344) | 0.51 (9.25)

6. Secondary Outcome: Change From Baseline Over Time in In-clinic Measured Mean Pulse Pressure
Time Frame: weeks 4, 8 and 12
Population: There was no information in the Case Report Form (CRF)
Arm/Group | T80/A5
Number analyzed (Participants) | 0

7. Secondary Outcome: DBP and SBP Control and Response Rates After 4, 8 and 12 Weeks of Treatment Using In-clinic BP Measurements
Description: DBP control is defined as DBP <90 mmHg or <80 mmHg in patients with diabetes or renal impairment. SBP control is defined as SBP <140 mmHg or <130 mmHg in patients with diabetes or renal impairment. DBP response is defined as DBP <90 mmHg or <80 mmHg in patients with diabetes or renal impairment or a reduction from baseline >=10mmHg. SBP response is defined as SBP<140 mmHg or <130 mmHg in patients with diabetes or renal impairment or a reduction from baseline >=15mmHg.
Time Frame: weeks 4, 8 and 12
Population: FAS and LOCF
Measure: Number; unit: Number of participants
Arm/Group | T80/A5
Number analyzed (Participants) | 494
Number of participants
  Week 4 DBP control | 313
  Week 8 DBP control | 368
  Week 12 DBP control | 373
  Week 4 SBP control | 247
  Week 8 SBP control | 305
  Week 12 SBP control | 311
  Week 4 DBP response | 329
  Week 8 DBP response | 393
  Week 12 DBP response | 399
  Week 4 SBP response | 337
  Week 8 SBP response | 388
  Week 12 SBP response | 393

8. Secondary Outcome: Percentage of Patients in Blood Pressure Categories Over Time
Description: BP optimal: SBP <120 mmHg and DBP <80 mmHg, BP normal: SBP <130 mmHg and DBP <85 mmHg but not optimal, BP high-normal: SBP <140 mmHg and DBP <90 mmHg but not normal. Grade 1 hypertension: SBP <160 mmHg and DBP <100 mmHg but not high-normal, Grade 2 hypertension: SBP <180 mmHg and DBP <110 mmHg but not grade 1, Grade 3 hypertension: SBP >=180 mmHg or DBP >=110 mmHg.
Time Frame: weeks 4, 8 and 12
Population: FAS with non-missing data
Measure: Number; unit: Percentage of participants
Arm/Group | T80/A5
Number analyzed (Participants) | 494
Percentage of participants
  BP optimal at week 4 (N=482) | 4.1
  BP normal at week 4 (N=482) | 19.7
  BP high-normal at week 4 (N=482) | 30.5
  Grade 1 hypertension at week 4 (N=482) | 39.0
  Grade 2 hypertension at week 4 (N=482) | 6.2
  Grade 3 hypertension at week 4 (N=482) | 0.4
  BP optimal at week 8 (N=487) | 5.5
  BP normal at week 8 (N=487) | 22.2
  BP high-normal at week 8 (N=487) | 40.0
  Grade 1 hypertension at week 8 (N=487) | 27.7
  Grade 2 hypertension at week 8 (N=487) | 4.3
  Grade 3 hypertension at week 8 (N=487) | 0.2
  BP optimal at week 12 (N=487) | 4.5
  BP normal at week 12 (N=487) | 28.5
  BP high-normal at week 12 (N=487) | 35.5
  Grade 1 hypertension at week 12 (N=487) | 27.1
  Grade 2 hypertension at week 12 (N=487) | 4.1
  Grade 3 hypertension at week 12 (N=487) | 0.2

9. Secondary Outcome: DBP and SBP Control and Response Rates Morning and Evening Over Time HBPM Measurements
Description: DBP control: DBP <85 mmHg, SBP control: SBP <135 mmHg, DBP response: DBP <85 mmHg or a reduction from baseline >=10 mmHg, SBP response: SBP <135 mmHg or a reduction from baseline >= 15 mmHg
Time Frame: weeks 4, 8 and 12
Population: FAS and LOCF and with at least one post baseline HBPM measurement
Measure: Number; unit: Number of participants
Arm/Group | T80/A5
Number analyzed (Participants) | 409
Number of participants
  DBP control morning at week 4 | 256
  DBP control morning at week 8 | 242
  DBP control morning at week 12 | 252
  DBP control evening at week 4 | 272
  DBP control evening at week 8 | 247
  DBP control evening at week 12 | 263
  SBP control morning at week 4 | 204
  SBP control morning at week 8 | 198
  SBP control morning at week 12 | 206
  SBP control evening at week 4 | 204
  SBP control evening at week 8 | 183
  SBP control evening at week 12 | 190
  DBP response morning at week 4 (N=354) | 256
  DBP response morning at week 8 (N=354) | 242
  DBP response morning at week 12 (N=354) | 252
  DBP response evening at week 4 (N=354) | 272
  DBP response evening at week 8 (N=354) | 247
  DBP response evening at week 12 (N=354) | 263
  SBP response morning at week 4 (N=299) | 204
  SBP response morning at week 8 (N=299) | 198
  SBP response morning at week 12 (N=299) | 206
  SBP response evening at week 4 (N=299) | 204
  SBP response evening at week 8 (N=299) | 183
  SBP response evening at week 12 (N=299) | 190

10. Secondary Outcome: Frequency of Patients Requiring Up-titration to Telmisartan 80mg Plus Amlodipine 10mg Combination (T80/A10) to Achieve Blood Pressure Control Over Time
Time Frame: weeks 4 and 8
Population: FAS
Measure: Number; unit: Number of participants
Arm/Group | T80/A5
Number analyzed (Participants) | 501
Number of participants
  Week 4 (n=482) | 186
  Week 8 (n=284) | 46

ADVERSE EVENTS:
Time Frame: 12 weeks: From drug administration until end of treatment plus one day.
Groups:
- T80/A10: Telmisartan 80 mg plus Amlodipine 10 mg once daily
Arm/Group | T80/A5 | T80/A10
Serious Adverse Events (participants affected / at risk) | 1/501 | 1/232
Other Adverse Events (participants affected / at risk) | 26/501 | 41/232
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | T80/A5 (N=501) | T80/A10 (N=232)
Duodenal ulcer (Gastrointestinal disorders) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | T80/A5 (N=501) | T80/A10 (N=232)
Oedema peripheral (General disorders) | 26 | 41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.